CLINICAL TRIAL: NCT00413491
Title: National Screening i Danmark Med MR-scanning af Brystet Kontra Klinisk Mammografi Hos Kvinder Der er bærere af Risikogivende BRCA1 Eller BRCA2 Mutationer
Brief Title: National Screening in Denmark With MR Versus Mammography and Ultrasound of Women With BRCA1 or BRCA2 Mutations
Acronym: MR BRCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Danish Breast Cancer Cooperative Group
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: DBCG07MRBRCA; DBCG07MRBRCA
Record Dates: First submitted 2006-12-14; First posted 2006-12-19 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2009-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; BRCA1 gene; BRCA2 gene; Magnetic Resonance Imaging; Mammography; Ultrasonography
MeSH Terms: conditions — Breast Neoplasms; Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (1):
- 1 (Experimental): Comparison of MR and mammography
  Interventions: Procedure: MR mammography; Procedure: MR

INTERVENTIONS:
Procedure: MR mammography — MR mammography
Procedure: MR — MR

SUMMARY:
The purpose of the study is to determine whether MR of the breast is a better screening tool than mammography combined with ultrasound of the breast in women with BRCA1 or BRCA2 gene mutations.

DETAILED DESCRIPTION:
Study type : Interventional Study design: Diagnostic,Prospective,Non Randomised,Blinded,Efficacy study

Further study details as provided by DBCG ( Danish Breast Cancer Cooperative Group):

Primary outcome measures:

Diagnostic outcome of a yearly screening with MR versus combined mammography and ultrasound of the breast measured by accuracy, sensitivity, specificity, positive and negative predictive values.

Secondary outcome measures:

Comparison of diagnostic outcome of MR versus combined mammography and ultrasound, in women with dense breast tissue compared with women with fatty breast tissue.

Comparison of the cancers found in women with BRCA gene mutations compared with the cancers found in the background population in respect of morphology, size, histological type, axillary lymph node status and grade.

Study start : January 2007. Expected completion 2010.

Women with BRCA gene mutations are more likely than others to develop the disease at a young age when breast density is higher than at older age.The tumours often are more rapidly developing with a short presymptomatic phase. These factors are known to reduce the effectiveness of screening with mammography and mammography seems to have a low sensitivity in women with BRCA gene mutations. Other studies have shown that more than 50% of the cancers appears as interval cancers between two mammography screening examinations and many have positive axillary nodes at the time of diagnosis.

Around 610 women are tested BRCA gene positive in Denmark in year 2006. These women are offered a yearly screening with mammography combined with ultrasound and a clinical examination. The trial will test whether this screening offer should be combined with or replaced by MR mammography.

ELIGIBILITY:
Inclusion Criteria:

* women tested positive of BRCA1 or BRCA2 gene mutations
* referred for screening
* aged 25 - 70 years

Exclusion Criteria:

* general contraindications for MR
* pregnant or lactating
* men
* bilateral mastectomy
* ongoing treatment with chemotherapy
* metastatic breast cancer
* previous breast surgery less than 6 months before MR
* previous radiation therapy of the breast less than 1 year before
* incapable of managing her own affairs

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic outcome of a yearly screening with MR versus combined mammography and ultrasound of the breast measured by accuracy, sensitivity, specificity, positive and negative predictive values. | 3 years

SECONDARY OUTCOMES:
Comparison of diagnostic outcome of MR versus combined mammography and ultrasound, in women with dense breast tissue compared with women with fatty breast tissue. | 3 years
Comparison of the cancers found in women with BRCA gene mutations compared with the cancers found in the background population in respect of morphology, size, histological type, axillary lymph node status and grade. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ilse Vejborg, MD, Principal Investigator — Danish Breast Cancer Cooperative Group
Locations (4):
- Denmark (4):
  - Department of Radiology,Copenhagen University Hospital Rigshospitalet, Copenhagen
  - Department of Radiology, Esbjerg Sygehus, Esbjerg
  - Department of Radiology, Sygehus Vendsyssel, Hjørring
  - Department of Radiology, Svendborg Sygehus, Svendborg